CLINICAL TRIAL: NCT07339488
Title: Efficacy and Safety of Combining Intestinal Low Dose Radiotherapy Plus Tislelizumab and Chemotherapy for Conversion of Borderline Resectable/Unresectable Esophageal Squamous Cell Carcinoma
Brief Title: Intestinal Low-Dose Radiotherapy Plus Immunochemotherapy for Conversion of Borderline Resectable/Unresectable Esophageal Squamous Cell Carcinoma
Acronym: ILDR-03
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chuangzhen Chen (Other)
Collaborators: BeOne Medicines (Industry)
Responsible Party: Sponsor-Investigator, Chuangzhen Chen, Director, Shantou University Medical College
Organization: Shantou University Medical College (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUMC-ILDR03
Record Dates: First submitted 2025-12-01; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Borderline Resectable Carcinoma; Unresectable Cancer; Esophageal Squamous Cell Carcinoma (ESCC); Immune Checkpoint Inhibitor; Chemotherapy; Radiotherapy; Tislelizumab
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Immune Checkpoint Inhibitors; Drug Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ILDR plus immunochemotherapy plus surgery (Experimental): 1Gy/1F ILDR + albumin-bound paclitaxel (3 cycles of 260 mg/m² on day 1), cisplatin (3 cycles of 75 mg/m² on day 1), and tislelizumab (3 cycles of 200 mg on day 1) + surgery
  Interventions: Radiation: Intestinal Low Dose Radiotherapy-1Gy; Drug: PD-1/PD-L1 inhibitors; Drug: Chemotherapy; Procedure: Surgery

INTERVENTIONS:
Radiation: Intestinal Low Dose Radiotherapy-1Gy — 1Gy ILDR will be administered to patients in a single fraction. The radiation treatment volume composes both the jejunum and ileum.
Drug: PD-1/PD-L1 inhibitors — 3 cycles of tislelizumab（200 mg D1 q3w）
Drug: Chemotherapy — 3 cycles of albumin-bound paclitaxel（260 mg/m2 D1 q3w）+ cisplatin（75 mg/m2 D1 q3w）
Procedure: Surgery — McKeown esophagectomy or laparoscopic-assisted McKeown esophagectomy is recommended, with either two-and-a-half-field lymphadenectomy or three-field lymph node dissection.

SUMMARY:
Esophageal cancer (EC) ranks among the leading malignant gastrointestinal tumors globally in terms of both incidence and mortality. Cases of EC in China account for over 50% of the global total, with squamous cell carcinoma being the primary pathological type. Locally advanced EC (LAEC), particularly cases where radical surgical resection is not feasible, exhibits high recurrence rates and low 5-year survival rates. However, studies have shown that patients with LAEC who undergo comprehensive treatment followed by surgery experience significantly prolonged survival and improved quality of life compared to those who do not receive surgical intervention.

Current conversion treatment regimens under investigation include: chemotherapy alone, chemoradiotherapy, immunotherapy combined with chemotherapy, and immunotherapy combined with chemoradiotherapy-each of these approaches has distinct advantages and limitations. Immunochemotherapy has emerged as a current research focus: it not only demonstrates significantly superior efficacy compared to chemotherapy alone but also exhibits lower cumulative toxicity than radiotherapy-combined conversion regimens, resulting in a more favorable overall benefit-risk ratio. As such, it represents the most promising conversion treatment strategy.

Retrospective and prospective clinical studies have shown that low-dose radiotherapy targeting the small intestine can enhance the anti-tumor response of immune checkpoint inhibitors (ICIs) in patients with advanced solid tumor, prolong their overall survival, and increase the incidence of the abscopal effect. Further mechanistic investigations have revealed that intestinal low-dose radiotherapy (ILDR) may augment the immune cancerous lethality by modulating the gut microbiota and their metabolic profiles.

Based on the findings from these preliminary studies, the current research plans to conduct a prospective phase II single-arm clinical trial to investigate the efficacy and safety of ILDR combined with immunochemotherapy as conversion therapy in patients with borderline resectable or unresectable esophageal squamous cell carcinoma (BR/UR ESCC). This research plans to enroll at least 39 evaluable cases or a total of 43 cases in two seperated stages, focusing on patients with thoracic BR/UR ESCC. Patients will receive a single fraction of ILDR with a mean dose of 1 Gy, concurrently with 3 cycles of albumin-bound paclitaxel (260 mg/m² on day 1), cisplatin (75 mg/m² on day 1), and tislelizumab (200 mg on day 1). The efficacy and safety of the treatment will be evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily enroll in this study, sign an informed consent form, and demonstrate good compliance.
2. Age ≥18 years and ≤75 years; both sexes are eligible.
3. ECOG performance status score of 0-1.
4. Pathologically confirmed esophageal squamous cell carcinoma (ESCC) prior to surgery.
5. Thoracic esophageal cancer.
6. Unresectable lesions, defined as: T4 stage; marginally resectable T3 stage (invading other organs, e.g., trachea, bronchus, or aorta not ruled out by imaging); presence or absence of unresectable lymph nodes or metastatic lymph nodes invading adjacent organs; presence or absence of supraclavicular lymph node metastasis; or clinically confirmed unresectable disease by the surgeon.
7. No prior history of anti-tumor treatment, including chemotherapy, hormonal therapy, radiotherapy, or immunotherapy.
8. Baseline laboratory requirements (within 7 days prior to enrollment):

   Hematology:
   1. Hb≥90 g/L (no transfusion within 14 days)
   2. NEUT ≥1.5×10⁹/L
   3. PLT ≥100×10⁹/L
   4. WBC≥3×10⁹/L

   Biochemistry:
   1. ALT and AST≤2.5×ULN
   2. TBIL≤1.5×ULN
   3. SCr≤1.5×ULN; or CrCl≥60 mL/min Coagulation: APTT, INR, and PT≤1.5×ULN Thyroid function: TSH≤ULN (if abnormal, FT3/FT4 levels should also be considered; eligible if FT3/FT4 are normal) Echocardiography: LVEF≥50%
9. Female subjects need to agree to use contraception during the study and for 6 months post-study; serum pregnancy test negative within 7 days prior to enrollment; non-lactating. Male subjects must agree to use contraception during the study and for 6 months post-study.
10. No psychological, familial, social, or geographical factors that may impair protocol adherence.
11. Other parameters meet general clinical trial enrollment criteria.
12. The subject or authorized representative has read, fully understands the patient information sheet, and signed the informed consent form.

Exclusion Criteria:

1. Patients with distant metastases other than supraclavicular lymph node metastases.
2. Presence or high risk of esophageal perforation.
3. Patients with contraindications to radiotherapy or immune checkpoint inhibitor (ICI) therapy.
4. Patients who previously experienced unacceptable toxicity after receiving ICI therapy.
5. Patients with a history of thoracoabdominal/pelvic radiotherapy within 6 months prior to enrollment.
6. Adverse reactions from prior anti-tumor treatment have not recovered to CTCAE v5.0 grade≤1 (excluding toxicities deemed by the investigator to pose no safety risk, such as fatigue or alopecia).
7. Subjects with active, uncontrolled systemic bacterial, viral, or fungal infections despite optimal treatment.
8. Respiratory depression, airway obstruction, or tissue hypoxia.
9. Severe cardiac disease (i.e., NYHA functional class II or higher).
10. Markedly abnormal liver or kidney function (i.e., indicators >3 times the upper limit of normal).
11. Active hepatitis B, hepatitis C, HIV, or syphilis.
12. Active brain disease or central nervous system/meningeal metastases with significant symptoms, or impaired decision-making capacity.
13. Hypersensitivity to drugs included in the trial.
14. Drug and/or alcohol abuse.
15. Pregnant or lactating women.
16. Concurrent participation in another therapeutic clinical trial.
17. Major surgical procedure within 30 days prior to enrollment.
18. Use of antibiotics, antifungals, antivirals, or antiparasitics within 4 weeks prior to registration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate | From postoperative day 0 up to 15 weeks postoperatively.
  The proportion of patients who, following conversion therapy, exhibit no residual invasive cancer cells in either the primary tumor site or regional lymph nodes upon pathological evaluation of surgical resection specimens, expressed as a percentage of the total treated population.

SECONDARY OUTCOMES:
Major Pathological Response (MPR) Rate | From postoperative day 0 up to 15 weeks postoperatively.
  MPR is defined as the proportion of patients with ≤10% residual viable tumor cells in surgical specimens following treatment. Pathological evaluation requires standardized sampling and separate assessment of lymph node metastases.
Objective Response Rate (ORR) | Baseline, every 6 weeks during conversion therapy, postoperation, every 4 months following the first postoperative assessment with a maximum duration of 12 months.
  Proportion of patients achieving complete response (CR) or partial response (PR) (sustained ≥4 weeks) per RECIST v1.1 and iRECIST criteria.
Disease Control Rate (DCR) | Baseline, every 6 weeks during conversion therapy, postoperation, every 4 months following the first postoperative assessment with a maximum duration of 12 months.
  DCR is defined as the proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD) post-treatment, as measured by RECIST 1.1 and iRECIST criteria.
Adverse Event Incidence Rate | Up to 12 months after surgery.
  The proportion of patients experiencing adverse events of any grade (graded according to CTCAE 6.0, Common Terminology Criteria for Adverse Events, grades 1-5) during treatment.
1-Year Disease-Free Survival Rate (1y-DFSR) | Up to 12 months after surgery.
  The 1y-DFSR is defined as the proportion of patients remaining in a disease-free state at 12 months from surgery completion. A disease-free state refers to the absence of tumor recurrence, metastasis, progression or death from any cause.
1-Year Overall Survival Rate (1y-OSR) | Up to 12 months after surgery.
  The 1y-OSR is defined as the proportion of patients who have not experienced all-cause death at 12 months following the initiation of treatment.
Surgical Conversion Rate | Up to 12 months after surgery.
  Defined as the proportion of initially unresectable patients who are converted to resectable status following treatment.
R0 Resection Rate | From postoperative day 0 up to 15 weeks postoperatively.
  Defined as the proportion of radical surgeries achieving microscopically negative margins (margin ≥1 mm).

OTHER OUTCOMES:
Peripheral Blood Immune Landscape | Baseline, and at a follow-up time point within 6 weeks after completion of conversion therapy but before surgical resection.
  Flow cytometry analysis is performed on peripheral blood samples.
Peripheral Blood Transcriptomics | Baseline, and at a follow-up time point within 6 weeks after completion of conversion therapy but before surgical resection.
  RNA sequencing is performed on peripheral blood samples.
Peripheral Blood Immune Receptor Repertoire | Baseline, and at a follow-up time point within 6 weeks after completion of conversion therapy but before surgical resection.
  TCR sequencing is performed on peripheral blood samples.
Serum Metabolomics | Baseline, and at a follow-up time point within 6 weeks after completion of conversion therapy but before surgical resection.
  The wide arrays of metabolites in peripheral blood samples are analyzed qualitatively and quantitatively.
Serum Cytokine Analysis | Baseline, and at a follow-up time point within 6 weeks after completion of conversion therapy but before surgical resection.
  The wide arrays of cytokines in peripheral blood samples are analyzed qualitatively and quantitatively.
Tissue Transcriptomics | Baseline, and at a follow-up time point within 6 weeks after completion of conversion therapy but before surgical resection.
  RNA sequencing is performed on tissue samples.
Tissue Immune Receptor Repertoire | Baseline, and at a follow-up time point within 6 weeks after completion of conversion therapy but before surgical resection.
  TCR sequencing is performed on tissue samples.
Tissue Immunohistochemistry | Baseline, and at a follow-up time point within 6 weeks after completion of conversion therapy but before surgical resection.
  Multi-marker fluorescent immunohistochemistry is performed on tissue samples.
Changes of Intestinal Flora | Baseline, and at a follow-up time point within 6 weeks after completion of conversion therapy but before surgical resection.
  Fecal samples are analyzed by metagenomics sequencing.
Fecal Metabolomics | Baseline, and at a follow-up time point within 6 weeks after completion of conversion therapy but before surgical resection.
  The wide arrays of metabolites in fecal samples are analyzed qualitatively and quantitatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Shantou University Medical College, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No